CLINICAL TRIAL: NCT02153554
Title: Capacity of State and Local Actors to Respond to Violence Against Women: Impact Evaluation of Training Civil Servants on Violence Against Women in Medellín (Colombia), Component of the Program "Seguridad Pública"
Brief Title: Impact Evaluation of Training Civil Servants on Violence Against Women in Medellín, Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Econometría Consultores (Other)
Collaborators: Inter-American Development Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATN/MG-13064-RG ECO 577-3
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Violence Against Women (VAW)

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Trained (Experimental): Training civil servants in Medellin (Colombia) on attention to violence against women.
  Interventions: Behavioral: Training civil servants on attention to violence against women
- Non trained (No Intervention)

INTERVENTIONS:
Behavioral: Training civil servants on attention to violence against women — The Secretary of Women of Medellin, through the ICONTEC, intends to conduct training to officials of the 22 family commissioners in Medellin. The objective of these trainings is to standardize procedures in order that women do not feel re-victimized and can forward complaints.
  Arms: Trained

SUMMARY:
The purpose of this study is to determine whether the training of civil servants leads to a reduction in the violence suffered by women, as well as in their psychological wellbeing and attitudes towards violence.

DETAILED DESCRIPTION:
The Secretary of Women of Medellin, through the ICONTEC, intends to conduct training to officials of the 22 family commissioners in Medellin. The objective of these trainings is to standardize procedures in order that women do not feel re-victimized and can forward complaints. Since the training will be done in phases in 2014 and there is willingness of relevant stakeholders to generate a random order on which commissioners the training is first performed, it can be done a cluster randomized trial.

We will require all 22 commissioners to be randomly assigned into two groups, one treatment and one control. To implement it is intended to:

* Conduct a baseline survey amongst women who used the services of the commissionaires between June and Septmber 2013, completed the process of care and signed informed consent.
* Training of a randomly chosen set of 11 commissioners will take place between June and September 2014.
* Conduct an endline survey amongst women who used the services of any of the 22 commissionaires between June and September 2014, completed the process of care and signed informed consent.

Women will be contacted through the commissioners. Women who have completed the process of care will be ask whether they want to participate in the study. If they agree, their contact details will transfer to the investigators for the survey to be conducted. This process would be conducted twice for baseline information before beginning the training, and for endline, once half of the first 11 commissioners have been trained.

ELIGIBILITY:
Inclusion Criteria:

* Women who initiate and finalize the process with the comissaries of family

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 975 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of violence | 3 months
  The outcome will be measure through a survey to women who used the services of the commissionaires, completed the process of care and signed informed consent

SECONDARY OUTCOMES:
Knowledge, attitudes and practices (KAP) on violence and care pathways | Average of 8 months after the complaint was presented at the comissaries
  The outcome will be measure through a survey to women who used the services of the commissionaires, completed the process of care and signed informed consent
Psychological well-being (self-acceptance, positive relationships, autonomy, environmental mastery, personal growth, purpose in life) | Average of 8 months after the complaint was presented at the comissaries
  The outcome will be measure through a survey to women who used the services of the commissionaires, completed the process of care and signed informed consent
Time resolution of cases | Average of 8 months after the complaint was presented at the comissaries
  The outcome will be measured through secondary data of the commissaries with information between the time of the initiation of the complaint and the completed the process of care.

CONTACTS AND LOCATIONS:
Locations (1):
- Econometria Consultores, Bogotá, Colombia